CLINICAL TRIAL: NCT00923234
Title: A Phase I Study of a Combination of 5-azacitidine Followed by Lenalidomide in High-risk MDS or Relapsed/Refractory AML Patients With Cytogenetic Abnormalities Including -5 or Del(5q)
Brief Title: Combination of 5-azacitidine and Lenalidomide in Myelodysplastic Syndromes (MDS) or Acute Myelogenous Leukemia (AML) Myelodysplastic Syndromes
Acronym: AZALE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The primary objective has already been answered with the number of recruited patients.
Sponsor: Technische Universität Dresden (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-AZALE1-037
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Myelodysplastic Syndromes; Acute Myelogenous Leukemia
Keywords: monosomy 5; del5q; lenalidomide; azacitidine
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine and Lenalidomide (Experimental): Azacitidine 75 mg/m² SC days 1-5 every 28 days for a maximum of 8 cycles and Lenalidomide 10 - 25 mg PO days 6-19 every 28 days for a maximum of 8 cycles
  Interventions: Drug: Azacitidine; Drug: Lenalidomide

INTERVENTIONS:
Drug: Azacitidine — 75 mg/m² SC days 1-5 every 28 days for a maximum of 8 cycles
  Other Names: Vidaza
Drug: Lenalidomide — 10 - 25 mg PO days 6-19 every 28 days for a maximum of 8 cycles
  Other Names: Revlimid

SUMMARY:
The hypothesis of this study is that 5-aza and lenalidomide act synergistically in MDS and AML patients with chromosomal abnormalities involving monosomy 5 or del5q. Therefore, this phase I study will investigate the maximum tolerated dose (MTD) of lenalidomide in combination with a fixed dose of 5-aza in this patient population.

DETAILED DESCRIPTION:
Cytogenetics are the main predictors of outcome in patients with AML. In fact, a monosomy 5 or del (5q) as single aberration are poor prognostic markers. Overall, the complete response rate for conventionally treated patients with newly-diagnosed AML with chromosome 5 abnormalities is about 31% to 37 % and all patients rapidly relapse if not rescued by allogeneic HSCT. The situation is almost similar in patients with high-risk MDS.Vidaza® has been shown in clinical trials to achieve remission rates in about 29% (CR+PR) of the patients while a total of 49% achieve improvement of blood counts.Revlimid® is also able to achieve complete remissions in advanced MDS and even overt leukemia with or without chromosome 5 abnormalities. Nevertheless, response rates are lower compared to low-risk MDS (IPSS Low/INT-1). Therefore, Revlimid® seems to be too weak as a single agent, but a promising compound for a combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age >=18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Relapsed or refractory AML (>30% blasts, FAB classification)with karyotype abnormalities involving monosomy 5 or del(5q) or MDS and t-MDS INT-2 or HIGH according to IPSS classification with karyotype abnormalities involving monosomy 5 or del(5q) either previously treated or untreated
* Not eligible for an immediate allogeneic HSCT (due to donor unavailability)
* All previous MDS or AML specific therapy with exception of corticosteroids not exceeding doses of 10mg/day prednisone must have been discontinued at least 1 week prior to study enrollment.
* Non-hematological toxicity (except alopecia) resulting from previous treatment must be resolved to WHO CTC Grade ≤ 2.
* ECOG performance status of < 3 at study entry.
* Laboratory test results within these ranges:Serum creatinine <= 2.0 mg/dL, Total bilirubin <= 3 x ULN, AST (SGOT) and ALT (SGPT) <= 3 x ULN
* Females of childbearing potential must agree to use a reliable form of contraception or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while on study).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Known hypersensitivity to thalidomide, lenalidomide, 5-azacitidine or mannitol.
* Myocardial infarction within 6 months before study entry, New York Heart Association Class III or IV heart failure, uncontrolled angina or severe uncontrolled ventricular arrhythmias.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Uncontrolled lung disease.
* Known positive for HIV or acute infectious hepatitis, type A, B or C.
* Participation in another clinical study in the 4 weeks prior to enrollment or during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Revlimid® (lenalidomide)in combination with Vidaza®(5-azacitidine) | during first cycle of therapy

SECONDARY OUTCOMES:
Clinical and cytogenetic response | during therapy
Safety (type, frequency, severity, and relationship of adverse events to study treatment) | during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, MD, Principal Investigator — Medizinische Klinik und Poliklinik I, Universitätsklinikum Carl Gustav Carus
Locations (4):
- Germany (4):
  - Medizinische Klinik und Poliklinik I, Uniklinik, Dresden
  - Universitätsklinikum Düsseldorf, Klinik für Hämatologie/Onkologie/klinische Immunologie, Düsseldorf
  - Klinikum der J.W. Goethe-Universität, Medizinische Klink II, Frankfurt
  - Technische Universität München, Klinikum Rechts der Isar, München